CLINICAL TRIAL: NCT03973502
Title: Application of 18F-FDOPA PET and Magnetic Resonance Spectroscopy (MRS) in Research of the Association Between HCV Infection and Parkinson's Disease.
Brief Title: Application of 18F-FDOPA PET and Magnetic Resonance Spectroscopy (MRS) With HCV and PD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201506041MINA
Record Dates: First submitted 2019-05-30; First posted 2019-06-04 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2022-05

CONDITIONS: Hepatitis C; Hepatitis B; Parkinson Disease
Keywords: Hepatitis C; Hepatitis B; Parkinson's disease; 18F-FDOPA PET, MRS; MRS
MeSH Terms: conditions — Hepatitis C; Hepatitis B; Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-DOPA PET (Experimental): PET/CT
  Interventions: Drug: 18F-DOPA PET

INTERVENTIONS:
Drug: 18F-DOPA PET — One hour later all patient will be injected intravenously with 185 MBq (5mCi) 18F-FDOPA. PET emission data acquisition in 3-dimensional mode will be started at 60 minutes after tracer injection for 30 minutes.

SUMMARY:
The objective of this study is to investigate the evidence of dopaminergic toxicity causing by HCV infection using 18F-FDOPA PET and MRS as imaging biomarkers.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the most common neurodegenerative disorder after Alzheimer's disease. It is characterized by degeneration of the dopaminergic neurons in substantia nigra and striatum, even before the clinical symptoms develop. Although the pathogenesis is still unclear, some viruses have been shown to be associated with acute or chronic parkinsonism. Recent studies have found that Hepatitis C virus (HCV) can replicate in the central nervous system, suggesting a possible link between PD and HCV. At the population and epidemiology level, the HCV infection and PD are strongly associated. At the molecular level, both HCV and PD have in common the overexpression of inflammatory biomarkers. Neuronal toxicity induced by HCV was also demonstrated. The positive association between HCV infection and PD has clinical implications for high endemic HCV areas, including Taiwan.

18F-FDOPA, an analog to L-DOPA, has been used as a positron-emitting compound for PET examination of patients affected by PD. It has been shown that putamen 18F-FDOPA uptakes are reduced by at least 35% at onset of symptoms, making the 18F-FDOPA PET as an imaging biomarker for detecting subclinical and preclinical parkinsonism. Earlier imaging study using magnetic resonance spectroscopy (MRS) to investigate cerebral effect of HCV also showed that chronic HCV infection had elevated choline/creatine ratios, a biomarker indicating inflammatory and infective conditions, in the basal ganglia and white matter.

The objective of this study is to investigate the evidence of dopaminergic toxicity causing by HCV infection using 18F-FDOPA PET and MRS as imaging biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Test Group

  1. Age：above 20 years old with HBV or HCV subjects.
  2. Patient agrees to participate in the study and receive UPDRS, MMSE, BDI II, MRI and PET imaging.
* Control Group

  1. Age：above 20 years old without carriers of Hepatitis B and C (ex. fatty liver), and no known neurological (ex. stroke, Parkinson's disease and degenerative neuropathy, etc.) and mental illness.
  2. Patient agrees to participate in the study and receive UPDRS, MMSE, BDI II, MRI and PET imaging.

Exclusion Criteria:

1. Patients could not receive PET and MRI studies, including panic mood to MRI study, allergy to contrast medium, hemodynamic instability.
2. Patients with pregnancy or recently having a plan for pregnancy.
3. Patient or family who does not agree to participate in the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2017-06-12 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
PET imaging | in 3 days
  Visual interpretation will be performed first by two independent readers to record if there is any abnormal 18F-FES accumulation. The presence, number, size, character, and location of suspected lesions will be filed for each patient in this study. The final results will be validated by tissue proof, correlation with other imaging, or follow-up results. Semi-quantitative analysis will be performed for each lesion suspected during visual interpretation. Standardized uptake values (SUV) will be obtained by placing regions of interest (ROIs) around the lesions that are identified on visual analysis. The maximum SUV (SUVmax) will be recorded.
  Volumetric parameters will be performed by placing volume of interests (VOIs) around the suspected lesions. VOIs will be generated using defined fix SUV thresholds or algorithm-generated isocontours. Manual adjustment of VOIs is allowed when non-tumoral tissue is incorrectly included by automatic method.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan